CLINICAL TRIAL: NCT03596151
Title: Clinical Study of a Single-Use, Point-of-Care Molecular Diagnostic Device for the Detection of Neisseria Gonorrhoeae (NG), Trichomonas Vaginalis (TV), and Chlamydia Trachomatis (CT) Utilizing Vaginal Swabs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: To optimize device
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0024; HHSN272201300014I
Record Dates: First submitted 2018-07-05; First posted 2018-07-23 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2018-06-22

CONDITIONS: Chlamydial Infection; Gonorrhoea; Trichomoniasis
Keywords: Chlamydia trachomatis; device; diagnostic; molecular; Neisseria gonorrhoeae; Trichomonas vaginalis
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Trichomonas Infections; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Click Device (Experimental): One self collected vaginal swab for Click Device testing. Three health care provider collected vaginal swabs for comparator testing.
  Interventions: Device: Click Device

INTERVENTIONS:
Device: Click Device — A single-use device containing a polymerase chain reaction (PCR)-based nucleic acid amplification test (NAAT) for detection of deoxyribonucleic acid (DNA) from Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), and Trichomonas vaginalis (TV) in self-collected vaginal specimens.

SUMMARY:
This is a multi-center study with a minimum of three sites in the United States. The study will enroll approximately 1750 female subjects and will have a study duration of approximately 9 months after enrollment of the first subject. Female subjects seen at the participating sites for any reason will be evaluated for enrollment in this study. All subjects will be managed per standard of care as applicable. Subjects who are enrolled in the study will perform self-collection of a vaginal swab to be tested by Click device, and allow the health care provider (HCP) to collect three additional vaginal swabs to be tested by recognized FDA-cleared comparator methods. Subjects will complete the study in a single visit. The primary objective is to assess the performance of the Click device for detection of Chlamydia trachomatis (CT), Neisseria gonorrhoeae (NG), and Trichomonas vaginalis (TV) in self-collected vaginal specimens as compared to Patient Infected Status (PIS) determined by three approved comparator assays using vaginal specimens collected by a qualified HCP in support of obtaining FDA clearance.

DETAILED DESCRIPTION:
This study is a multi-center study with a minimum of three Clinical Laboratory Improvement Amendments-waived (CLIA-waived) intended operator sites in the United States; approximately one-third of the total number of sites will have a patient population of low Neisseria gonorrhoeae (NG), Chlamydia trachomatis (CT), or Trichomonas vaginalis (TV) prevalence. Low prevalence sites are defined as sites with a prevalence < / = 2% for any of the three targets. Sites with a prevalence higher than 2% for any of the three targets will be defined as high prevalence sites. The study will enroll approximately 1750 female subjects and will have a study duration of approximately 9 months after enrollment of the first subject. Approximately one-third of the total subjects shall be recruited from low prevalence sites for the infections of interest. Female subjects seen at the participating sites for any reason will be evaluated for enrollment in this study. All subjects will be managed per standard of care as applicable. Subjects who are enrolled in the study will perform self-collection of a vaginal swab to be tested by Click device, and allow the health care provider (HCP) to collect three additional vaginal swabs to be tested by recognized FDA-cleared comparator methods. Subjects will complete the study in a single visit. The hypothesis of this study is that the identification of each organism (CT, NG, and TV) in self-collected vaginal swabs by women using the Click device will agree with the Patient Infected Status (PIS) with a high sensitivity and specificity. The primary objective is to assess the performance of the Click device for detection of CT, NG, and TV in self-collected vaginal specimens as compared to PIS determined by three approved comparator assays using vaginal specimens collected by a qualified HCP in support of obtaining FDA clearance. The secondary objectives are: 1) to assess the performance of the Click device for detection of CT, NG, and TV in self-collected vaginal specimens among symptomatic subjects as compared to PIS determined by three approved comparator assays using vaginal specimens collected by a qualified HCP; 2) to assess the performance of the Click device for detection of CT, NG, and TV in self-collected vaginal specimens among asymptomatic subjects as compared to PIS determined by three approved comparator assays using vaginal specimens collected by a qualified HCP.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give voluntary written informed consent (or the parent/legal guardian will provide parental permission) before any study-related procedure is performed.
2. Female at birth. (Pregnant and breastfeeding women are eligible)
3. Age > / = 14 years at the time of enrollment.
4. Able to read and understand the procedural information provided for the study.
5. Able and willing to follow all study procedures, including performing self-collection of one vaginal swab and permitting a licensed health care provider to collect three additional vaginal swabs.

Exclusion Criteria:

1. Have a medical condition, serious intercurrent illness, or other circumstance that, in the Investigator's judgment, could jeopardize the subject's safety, or could interfere with study procedures.
2. Enrollment in this study previously.

Ages: 14 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Axis Clinical Trials, Los Angeles, California
  - University of California, San Diego - Antiviral Research Center, San Diego, California
  - San Francisco Department of Public Health - San Francisco City Clinic, San Francisco, California
  - Florida International University - Student Health Center, Miami, Florida
  - Cook County Health and Hospitals System - Ruth M Rothstein CORE Center, Chicago, Illinois
  - Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland
  - University of Mississippi - Infectious Diseases, Jackson, Mississippi
  - Magee Women's Hospital of UPMC - Reproductive Infectious Disease Research, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Click Device: The study population was comprised of female participants >=14 years of age who visited any of the participating clinics for any reason, who may have been symptomatic or asymptomatic for STIs at locations including but not limited to: OB/GYN and primary care offices, as well as sexually transmitted disease, teen, public health, and family planning clinics.
  Participants who met the inclusion/exclusion criteria were offered enrollment into the study. Participants who enrolled in the study provided clinical and demographic information, performed self-collection with a vaginal swab for the Click device, and allowed the health care professional (HCP) to collect three additional vaginal swabs for the comparator methods. Participants completed the study in a single visit.
Period: Overall Study
Arm/Group | Click Device
Started | 295
Completed | 294
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants who were enrolled in the study.
Groups:
- Click Device: The study population was comprised of female participants >=14 years of age who visited any of the participating clinics for any reason, who performed self-collection with a vaginal swab for the Click device, and allowed the health care professional (HCP) to collect three additional vaginal swabs for the comparator methods.
Arm/Group | Click Device
Number analyzed (Participants) | 295
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 286
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 194
  Unknown or Not Reported | 77
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 13
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 151
  White | 80
  More than one race | 23
  Unknown or Not Reported | 25
Region of Enrollment [Number; unit: participants]
  United States | 295
Symptomatic Status [Count of Participants; unit: Participants]
  Symptomatic | 168
  Asymptomatic | 127
Evaluable for NG [Count of Participants; unit: Participants] — Population: Participants who are deemed evaluable for Neisseria gonorrhoeae (NG).
  Participants
    number analyzed (Participants) | 255
    Symptomatic | 149
    Asymptomatic | 106
Evaluable for CT [Count of Participants; unit: Participants] — Population: Participants who are deemed evaluable for Chlamydia trachomatis (CT).
  Participants
    number analyzed (Participants) | 256
    Symptomatic | 149
    Asymptomatic | 107
Evaluable for TV [Count of Participants; unit: Participants] — Population: Participants who are deemed evaluable for Trichomonas vaginalis (TV).
  Participants
    number analyzed (Participants) | 255
    Symptomatic | 148
    Asymptomatic | 107

OUTCOME MEASURES:

1. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device for Detection of Chlamydia Trachomatis (CT) in Self-collected Vaginal Specimens as Compared to Patient Infection Status (PIS) Using Vaginal Specimens Collected by a Qualified HCP
Description: The sensitivity of the Click device is defined as follows:
  TP = the number of specimens where both the Click result and the PIS designation are Positive; FN = the number of specimens where the Click result is Negative and the PIS designation is Positive; Sensitivity = 100 * TP / (TP + FN)
  The specificity of the Click device is defined as follows:
  TN = the number of specimens where both the Click result and the PIS designation are Negative; FP = the number of specimens where the Click result is Positive and the PIS designation is Negative; Specificity = 100 * TN / (TN + FP)
Time Frame: Day 1
Population: This population includes all participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for CT. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result.
Measure: Count of Participants; unit: Participants
Groups:
- Click Device: The study population was comprised female participants >=14 years of age who visited any of the participating clinics for any reason, who performed self-collection with a vaginal swab for the Click device, and allowed the health care professional (HCP) to collect three additional vaginal swabs for the comparator methods.
Arm/Group | Click Device
Number analyzed (Participants) | 256
Participants
  Sensitivity: number analyzed (Participants) | 10
  Sensitivity | 10
  Specificity: number analyzed (Participants) | 246
  Specificity | 241

2. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device for Detection of Neisseria Gonorrhoeae (NG) in Self-collected Vaginal Specimens as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP
Description: as for outcome 1
Time Frame: Day 1
Population: This population includes all participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for NG. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result.
Measure: Count of Participants; unit: Participants
Arm/Group | Click Device
Number analyzed (Participants) | 255
Participants
  Sensitivity: number analyzed (Participants) | 0
  Sensitivity | 0
  Specificity | 249

3. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device for Detection of Trichomonas Vaginalis (TV) in Self-collected Vaginal Specimens as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP
Description: as for outcome 1
Time Frame: Day 1
Population: This population includes all participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for TV. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result.
Measure: Count of Participants; unit: Participants
Arm/Group | Click Device
Number analyzed (Participants) | 255
Participants
  Sensitivity: number analyzed (Participants) | 30
  Sensitivity | 29
  Specificity: number analyzed (Participants) | 225
  Specificity | 212

4. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of CT as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP Among Symptomatic Participants
Description: as for outcome 1
Time Frame: Day 1
Population: This population includes all symptomatic participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for CT. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result. If a participant reported "Yes" to any of the symptoms on the Clinical Symptoms Assessment form, the participant is classified as Symptomatic. Otherwise, the participant is classified as "Asymptomatic".
Measure: Count of Participants; unit: Participants
Arm/Group | Click Device
Number analyzed (Participants) | 149
Participants
  Sensitivity: number analyzed (Participants) | 6
  Sensitivity | 6
  Specificity: number analyzed (Participants) | 143
  Specificity | 139

5. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of NG as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP Among Symptomatic Participants
Description: as for outcome 1
Time Frame: Day 1
Population: This population includes all symptomatic participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for NG. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result. If a participant reported "Yes" to any of the symptoms on the Clinical Symptoms Assessment form, the participant is classified as Symptomatic. Otherwise, the participant is classified as "Asymptomatic".
Measure: Count of Participants; unit: Participants
Arm/Group | Click Device
Number analyzed (Participants) | 149
Participants
  Sensitivity: number analyzed (Participants) | 0
  Sensitivity | 0
  Specificity | 145

6. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of TV as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP Among Symptomatic Participants
Description: as for outcome 1
Time Frame: Day 1
Population: This population includes all symptomatic participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for TV. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result. If a participant reported "Yes" to any of the symptoms on the Clinical Symptoms Assessment form, the participant is classified as Symptomatic. Otherwise, the participant is classified as "Asymptomatic".
Measure: Count of Participants; unit: Participants
Arm/Group | Click Device
Number analyzed (Participants) | 148
Participants
  Sensitivity: number analyzed (Participants) | 17
  Sensitivity | 17
  Specificity: number analyzed (Participants) | 131
  Specificity | 124

7. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of CT as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP Among Asymptomatic Participants
Description: as for outcome 1
Time Frame: Day 1
Population: This population includes all asymptomatic participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for CT. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result. If a participant reported "Yes" to any of the symptoms on the Clinical Symptoms Assessment form, the participant is classified as Symptomatic. Otherwise, the participant is classified as "Asymptomatic".
Measure: Count of Participants; unit: Participants
Arm/Group | Click Device
Number analyzed (Participants) | 107
Participants
  Sensitivity: number analyzed (Participants) | 4
  Sensitivity | 4
  Specificity: number analyzed (Participants) | 103
  Specificity | 102

8. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of NG as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP Among Asymptomatic Participants.
Description: as for outcome 1
Time Frame: Day 1
Population: This population includes all asymptomatic participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for NG. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result. If a participant reported "Yes" to any of the symptoms on the Clinical Symptoms Assessment form, the participant is classified as Symptomatic. Otherwise, the participant is classified as "Asymptomatic".
Measure: Count of Participants; unit: Participants
Arm/Group | Click Device
Number analyzed (Participants) | 106
Participants
  Sensitivity: number analyzed (Participants) | 0
  Sensitivity | 0
  Specificity | 104

9. Primary Outcome: The Percent Sensitivity and Percent Specificity of Click Device Using Self-collected Vaginal Swabs for Detection of TV as Compared to PIS Using Vaginal Specimens Collected by a Qualified HCP Among Asymptomatic Participants.
Description: as for outcome 1
Time Frame: Day 1
Population: This population includes all asymptomatic participants with samples that provide an evaluable Click Diagnostics Sexual Health Test result and an evaluable PIS result for TV. An evaluable result is indicated if both the Click device and the PIS provide a valid positive or negative result. If a participant reported "Yes" to any of the symptoms on the Clinical Symptoms Assessment form, the participant is classified as Symptomatic. Otherwise, the participant is classified as "Asymptomatic".
Measure: Count of Participants; unit: Participants
Arm/Group | Click Device
Number analyzed (Participants) | 107
Participants
  Sensitivity: number analyzed (Participants) | 13
  Sensitivity | 12
  Specificity: number analyzed (Participants) | 94
  Specificity | 88

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Click Device
All-Cause Mortality (participants affected / at risk) | 0/294
Serious Adverse Events (participants affected / at risk) | 0/294
Other Adverse Events (participants affected / at risk) | 0/294

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03596151/Prot_SAP_000.pdf